CLINICAL TRIAL: NCT01662180
Title: Predicting Ovarian Response in Artificial Insemination With Low Stimulation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Isala (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Principal Investigator, M. Bloemendal, drs., Isala
Other Study IDs: PRORAILS trial
Record Dates: First submitted 2012-07-26; First posted 2012-08-10 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Subfertility
Keywords: subfertility, IUI, rec FSH, FSH, E2, AMH
MeSH Terms: conditions — Infertility | interventions — Follicle Stimulating Hormone; follitropin beta; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample tested for FSH, E2 and AMH
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subfertile couples: Subfertile couples presenting at fertility clinics with an indication for IUI in stimulated cycles
  All patients will receive a fixed 75 IU recombinant follicle stimulating hormone per day conform normal stimulation protocol starting from cycle day 3, 4 or 5. Once the dominant follicle(s) reach a mean diameter of 16-18 mm, hCG (5000IU or 250 mcg) will be applied and insemination will be scheduled 36-42 hours later. Patients will be followed for the time of one menstrual cycle.
  Interventions: Drug: Follicle Stimulating Hormone

INTERVENTIONS:
Drug: Follicle Stimulating Hormone — All patients will receive a fixed 75 IU rec follicle stimulating hormone per day subcutaneous injection stimulation protocol starting from cycle day 3, 4 or 5. The intervention done in this study is conform normal stimulation protocol and is not the target of this study.
  Other Names: Puregon [Merck Sharp & Dohme bv]; Gonal -F [Serono Benelux bv]

SUMMARY:
This large prospective multi-center cohort study aims to identify patient's characteristics that significantly influence ovarian response to mild stimulation with a fixed dose of 75 IU recombinant FSH.

DETAILED DESCRIPTION:
A multi-center, open-label, prospective cohorts study. Patients with a regular indication for COH/IUI (controlled ovarian stimulation/ intra uterine insemination) will be asked to participate. Patient's characteristics will be documented including age, weight, BMI, smoking status, cycle day 2 3 or 4 FSH /Estradiol levels, antral follicle count, and AMH. AMH and FSH/Estradiol will be determined centrally after completion of inclusion of all patients in the study. All patients will receive a fixed 75 IU recFSH per day conform normal stimulation protocol starting from cycle day 3, 4 or 5 after exclusion of ovarian cysts by ultrasound. Ovarian response will be documented by ultrasound only. Once the dominant follicle(s) reach a mean diameter of 16-18 mm, hCG (5000IU or 250 mcg) will be applied and insemination will be scheduled 36-42 hours later. Cancellation criteria will be defined according to the national guidelines provided by the NVOG (7).

ELIGIBILITY:
Inclusion Criteria:

* couples with unexplained or mild male subfertility (1-3) and a spontaneous chance of conception below 40% (Hunault score).
* Unexplained subfertility including minimal to mild endometriosis (AFS grade 1 or 2) is defined as the failure to conceive after at least one year of unprotected intercourse whereas the standard fertility work-up was unable to detect any factors that might influence fertility negatively.
* semen analysis should be normal according to the WHO guidelines (8),
* ovulation should be documented (by BBT charts, ovulation detection by ultrasound or normal luteal progesterone values),
* tubal patency should be confirmed (HSG, laparoscopy or fertiloscopy) and when a postcoital test was performed a cervical factor should have been excluded.
* Mild male subfertility is defined as abnormal semen parameters according to the WHO (8) but an average total motile sperm account before processing of at least 10 million.

Exclusion Criteria:

* Hunault score ≥ 40%
* Endometriosis AFS grade 3 or 4
* Contra-indications for the use of gonadotrophins (cysts larger than 2 cm, allergy for gonadotrophins)
* Total motile sperm count after sperm processing below 1 million
* Women aged younger than eighteen years or older than 45 years.
* Previous treatment with COH/IUI for treating current subfertility
* Unable to speak or read the Dutch language

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subfertile couples presenting at fertility clinics with an indication for IUI in stimulated cycles
Sampling Method: Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-09 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
To assess the relationship between AMH serum levels and ovarian response | one menstrual cycle, one month
  (defined by the number of dominant follicles >15mm) in IUI cycles stimulated with a fixed dose of 75 IU recFSH. All follicles > 11 mm will be documented

SECONDARY OUTCOMES:
To assess the relationship between age, weight, BMI, smoking, AFC, FSH/E2 on CD3 and ovarian response | one menstrual cycle, one month
  (defined by the number of dominant follicles >15mm) in IUI cycles stimulated with a fixed dose of 75 IU recFSH.
Pregnancy rate per started cycle. | three months
  From start of the menstrual cycle until a positive heartbeat registered at 12 weeks of gestation.
Multiple pregnancy rate per started cycle. | three months
  From start of the menstrual cycle until positive heartbeats registered at 12 weeks of gestation.
Miscarriage rate per started cycle. | five months
  miscarriage up to 16 weeks of gestation
Cancellation rate per stimulated cycle | one menstrual cycle, one month

CONTACTS AND LOCATIONS:
Overall Officials: Ben Cohlen, dr., Principal Investigator — Isala
Locations (7):
- Netherlands (7):
  - OLVG, Amsterdam, Po 95500
  - Isala Klinieken, Zwolle, PO Box 10400
  - Catharina Ziekenhuis, Eindhoven, PO Box 1350
  - AMC, Amsterdam, PO Box 22660
  - VUMC, Amsterdam, PO Box 7057
  - UMC Utrecht, Utrecht, PO Box 85500
  - st Elizabeth Gasthuis, Tilburg, PO Box 90151

REFERENCES:
- [Background] Bensdorp AJ, Cohlen BJ, Heineman MJ, Vandekerckhove P. Intra-uterine insemination for male subfertility. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD000360. doi: 10.1002/14651858.CD000360.pub4. PMID 17943739
- [Background] Verhulst SM, Cohlen BJ, Hughes E, Te Velde E, Heineman MJ. Intra-uterine insemination for unexplained subfertility. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD001838. doi: 10.1002/14651858.CD001838.pub3. PMID 17054143
- [Background] Tummon IS, Asher LJ, Martin JS, Tulandi T. Randomized controlled trial of superovulation and insemination for infertility associated with minimal or mild endometriosis. Fertil Steril. 1997 Jul;68(1):8-12. doi: 10.1016/s0015-0282(97)81467-7. PMID 9207576
- [Background] Freiesleben NL, Lossl K, Bogstad J, Bredkjaer HE, Toft B, Loft A, Bangsboll S, Pinborg A, Budtz-Jorgensen E, Andersen AN. Predictors of ovarian response in intrauterine insemination patients and development of a dosage nomogram. Reprod Biomed Online. 2008 Nov;17(5):632-41. doi: 10.1016/s1472-6483(10)60310-0. PMID 18983747
- [Background] la Cour Freiesleben N, Lossl K, Bogstad J, Bredkjaer HE, Toft B, Rosendahl M, Loft A, Bangsboll S, Pinborg A, Nyboe Andersen A. Individual versus standard dose of rFSH in a mild stimulation protocol for intrauterine insemination: a randomized study. Hum Reprod. 2009 Oct;24(10):2523-30. doi: 10.1093/humrep/dep239. Epub 2009 Jul 14. PMID 19602518
- [Background] Freiesleben Nl, Rosendahl M, Johannsen TH, Lossl K, Loft A, Bangsboll S, Friis-Hansen L, Pinborg A, Andersen AN. Prospective investigation of serum anti-Mullerian hormone concentration in ovulatory intrauterine insemination patients: a preliminary study. Reprod Biomed Online. 2010 May;20(5):582-7. doi: 10.1016/j.rbmo.2010.02.007. Epub 2010 Feb 12. PMID 20303323
- [Background] Cooper TG, Noonan E, von Eckardstein S, Auger J, Baker HW, Behre HM, Haugen TB, Kruger T, Wang C, Mbizvo MT, Vogelsong KM. World Health Organization reference values for human semen characteristics. Hum Reprod Update. 2010 May-Jun;16(3):231-45. doi: 10.1093/humupd/dmp048. Epub 2009 Nov 24. PMID 19934213
- [Background] La Marca A, Sighinolfi G, Radi D, Argento C, Baraldi E, Artenisio AC, Stabile G, Volpe A. Anti-Mullerian hormone (AMH) as a predictive marker in assisted reproductive technology (ART). Hum Reprod Update. 2010 Mar-Apr;16(2):113-30. doi: 10.1093/humupd/dmp036. Epub 2009 Sep 30. PMID 19793843
- [Background] Nelson SM, Anderson RA, Broekmans FJ, Raine-Fenning N, Fleming R, La Marca A. Anti-Mullerian hormone: clairvoyance or crystal clear? Hum Reprod. 2012 Mar;27(3):631-6. doi: 10.1093/humrep/der446. Epub 2012 Jan 11. PMID 22238112
- [Derived] Rutten A, van Ballegooijen H, Broekmans F, Cohlen B; PRORAILS study group. Insights into ovarian response with a fixed low dose FSH stimulation in an IUI programme: the PRORAILS study. Hum Reprod. 2022 Jun 30;37(7):1440-1450. doi: 10.1093/humrep/deac076. PMID 35460412